CLINICAL TRIAL: NCT07333300
Title: Exploratory Clinical Investigation on Neurosensory Responses Via EEG Headband in Adults With Mild to Moderate Atopic Dermatitis After Application of Marketed Product Compared With Placebo (Water Application).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NB250043-NB-V_1.0_16Oct25
Record Dates: First submitted 2025-11-15; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD)
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Test Product- CeraVe Moisturizing Lotion (Experimental): Arm 1 (Test Product): Subjects in this group will receive the marketed product, applied topically as per the study procedure.
  Interventions: Other: Marketed Test Product
- Placebo Comparator: Arm 2 (Experimental): Arm 2 (Placebo Control): Subjects in this group will receive a placebo (water application), in which no active ingredient will be added. The placebo will be identical in appearance and texture to the test product to maintain blinding.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Marketed Test Product — Topical Application Frequency: Single Application. Spread the cream in the same direction and avoid scratching after application.
  Arms: Arm 1 - Test Product- CeraVe Moisturizing Lotion
Other: Placebo — Topical Application Frequency : Single Application Spread the cream in the same direction and avoid scratching after application.
  Arms: Placebo Comparator: Arm 2

SUMMARY:
This is a prospective, exploratory, double-blind, single-visit internal validation study designed to evaluate neurosensory responses using electroencephalography head band (EEG) in adult subjects with mild to moderate atopic dermatitis (AD) following a single topical application of marketed product compared with placebo (water application).

DETAILED DESCRIPTION:
A total of twenty (20) subjects will be enrolled with ten in each arm, aged between 18 to 65 years, with mild to moderate AD for at least six months. Participants will be recruited after providing with the written subject information sheet, and eligibility will be determined based on predefined inclusion and exclusion criteria. The study consists of a single visit (Day 01), during which participants will undergo screening, randomization, enrolment, and baseline evaluations, followed by product application and post-application assessments up to 30 minutes, after which end-of-study procedures will be completed. Validation assessments will consist of EEG recordings to evaluate neurosensory responses in subjects with atopic dermatitis. The analysis will focus on changes in alpha, beta, and theta brainwave activity, which are key indicators of cortical processing related to sensory perception. In addition to EEG, digital photographs will be captured using a Nikon D3300 camera to document any visible skin changes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years (both inclusive) at the time of consent having mild to moderate atopic dermatitis. 2. Sex: Healthy male and non-pregnant/non-lactating females. 3. Females of childbearing potential must have a self-reported negative pregnancy test. 4. Subject are generally in good health. 5. Subjects who agree to come to the facility with clean and dry scalp and hair 6. Subjects with mild to moderate Atopic Dermatitis determined by Eczema

Area and Severity Index (EASI) score with moderate erythema (redness:

score 2) and mild scratch mark (scratching: score 1) will be enrolled into the study 7. Subjects are not allowed to participate in any other study until this study is complete. 8. Subjects willing and able to follow the study directions. 9. Having childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/ injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam,partner vasectomy or abstinence). Females will be considered as nonchildbearing potential if they are surgically sterile, have been postmenopausal for at least 1 year or have had a tubal ligation. 10. Subjects willing to give written consent through subject information sheet. 11. Subjects have not participated in a similar investigation in the past three months. 12. Subjects willing to use test product throughout the study period.

Exclusion Criteria:

* History of any dermatological condition of the skin diseases. 2. Subject with present condition of allergic response to any cosmetic product. 3. Subjects with other dermatologic diseases besides AD whose presence or treatments could interfere with the assessment of disease (eg, Psoriasis). 4. Subjects who used systemic immunosuppressants within 4 weeks, topical steroids or immunomodulators within 1 week, moisturizers within 12 hours before evaluation. 5. History of alcohol or drug addiction. 6. The subject has a known allergy or sensitivity to soaps, lotions, detergents, detanglers or fragrances. 7. The subject has any other skin conditions i.e. cuts, scratches, ring worms, etc. which in the opinion of the Investigator, will interfere with the study results or will create undue risk for the subject. 8. Subjects having diabetes, hepatitis, epilepsy, thyroid or have or had any kind of cancer. 9. The subject must not have participated in a clinical study within 4 weeks prior to the screening visit of this study. 10. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion. 11. Pregnant or breastfeeding or planning to become pregnant during the study period. 12. History of chronic illness which may influence the cutaneous state.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
To measure neurosensory responses associated with pain, pruritus, and discomfort in subjects with atopic dermatitis. | • Baseline (before application of the test product) • During Stimulus Induction • Post-stimulus induction (test product use) at T-30 minutes.
  To measure the changes in the
  * Alpha Wavelength activity
  * Beta Wavelength activity
  * Theta Wavelength activity It will be measured through MUSE Biosensing Headband. The headband will be applied over the subjects in head area and the electrodes will help in detection of the wavelength.

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Study Director — NovoBliss Research Private Limited

IPD SHARING:
Plan to Share IPD: No